CLINICAL TRIAL: NCT00296049
Title: An Open-Label, Pilot Study of Daptomycin vs. Vancomycin for Treatment of Gram-Positive Bacteremia in Neutropenic Cancer Patients
Brief Title: Daptomycin or Vancomycin in Treating Bacteria in the Blood in Patients With Neutropenia Caused By Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000466308; CCCWFU-98804; CUBIST-CCCWFU-98804; CCCWFU-BG04-494
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Infection; Neutropenia; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; infection; neutropenia; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Infections; Neutropenia | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vancomycin (Active Comparator)
  Interventions: Drug: vancomycin
- daptomycin (Experimental)
  Interventions: Drug: daptomycin

INTERVENTIONS:
Drug: daptomycin
  Arms: daptomycin
Drug: vancomycin
  Arms: vancomycin

SUMMARY:
RATIONALE: Antibiotics, such as daptomycin and vancomycin, may be effective in treating bacteria in the blood. It is not yet known whether daptomycin is more effective than vancomycin in treating bacteria in the blood in patients with neutropenia caused by chemotherapy.

PURPOSE: This randomized clinical trial is studying daptomycin to see how well it works compared with vancomycin in treating bacteria in the blood in patients with neutropenia caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety of daptomycin vs vancomycin in cancer patients with chemotherapy-induced neutropenia and gram-positive bacteremia.
* Compare the efficacy of these drugs, in terms of fever resolution, bacteremia resolution, inflammation indicators reduction, implanted catheter salvage, and reduced need for antifungal therapy, in these patients.

OUTLINE: This is an open-label, randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive daptomycin IV over 30 minutes once daily.
* Arm II: Patients receive vancomycin IV over 60 minutes twice daily. Treatment in both arms continues for approximately 7-14 days or until microbiologic failure, unsatisfactory clinical (symptomatic) response, or fever and neutropenia is resolved (absolute neutrophil count ≥ 1,000/mm^3 on ≥ 2 consecutive days). Patients may be removed from the study if the isolate is found to be sensitive to the original antibiotics or resistant to either of the study drugs.

After completion of study therapy, patients are followed at 6 and 12 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignancy
* Chemotherapy-induced neutropenia (absolute neutrophil count < 500/mm^3)
* Two or more blood cultures positive for gram-positive cocci

  * At least 0.2 colony-forming units/mL on lysis-centrifugation culture
* Currently receiving broad-spectrum antimicrobial therapy appropriate for febrile neutropenia
* No meningitis, endocarditis, osteomyelitis, or pneumonia (by clinical or radiologic criteria)

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 7 days
* No allergy or intolerance to vancomycin or daptomycin
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after completion of study treatment
* No underlying myopathy or neurologic disease (e.g., Guillan-Barre or multiple sclerosis)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent HMG CoA reductase inhibitors (statins)
* No concurrent gemfibrozil or clofibrate

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
determine the efficacy of daptomycin to treat gram positive infections | day 7
determine the safety of daptomycin in neutropenic patients | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Kevin High, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States